CLINICAL TRIAL: NCT01112215
Title: Randomized Controlled Trial to Evaluate the Efficacy of Enteric-coated Mycophenolate Sodium Versus Azathioprine for the Induction and Maintenance of Remission of the Extra-renal Lupus Manifestations
Brief Title: Enteric-coated Mycophenolate Sodium Versus Azathioprine for the Extra-renal Lupus Manifestations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008-008934-35
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2015-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; non-renal manifestations
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azathioprine (Active Comparator)
  Interventions: Drug: Azathioprine
- Enteric-coated Mycophenolate Sodium (Active Comparator)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium

INTERVENTIONS:
Drug: Azathioprine — Initial dose of 2-2.5 mg/kg (according to TMTP levels) for 6 months according the severity of the flare with progressive tapering if complete remission has been obtained
  Arms: azathioprine
Drug: Enteric-Coated Mycophenolate Sodium — Initial dose of 1440 mg/day for 6 months to be tapered progressively if complete remission had been obtained
  Arms: Enteric-coated Mycophenolate Sodium

SUMMARY:
Azathioprine is still considered the treatment of choice for the non-renal manifestations of systemic lupus erythematosus (SLE) with an estimated efficacy of 45%.Recently, several studies have demonstrated the efficacy of mycophenolate mofetil/enteric-coated mycophenolate sodium in those cases, but so far, no controlled, randomized comparative study between the two drugs has been conducted. The aim is to perform a randomized, controlled, phase III/IV study comparing enteric-coated mycophenolate (ECMs) with azathioprine for induction and maintenance therapy of the non-renal manifestations of SLE. Methods: Patients with non-renal SLE flares (SLEDAI≥6 and/or BILAG o 2B refractory to full doses of hydroxychloroquine and prednisolone (≥10 mg/d) or with relapsing flares will be included. Patients will be stratified according the flare severity (moderate (SLEDAI<12)-severe (SLEDAI≥12)) and randomized (1:1) into two groups of treatment, EMCs (2gr/d) or AZA (2-2.5mg/kg/d) according to TMPT levels for 6 months. Dose will be progressively tapered based on clinical response up to completing a year of treatment. The main aim is the percentage of complete remission achieved ((SLEDAI <4 and/or absence of any BILAG A o B) at week 12 and 24 for moderate and severe flares, respectively. Secondary objectives include evaluating the reduction in the steroid requirement, number of flares post-treatment, effect on the biological parameters, and impact on quality of life, damage and drug safety. To detect a 20% difference between the two drugs with a 80% statistical power (0.05 alpha error), considering a follow up loss of 20%, a total of 240 patients is required.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Fulfill at least 4 of the 11 criteria for the ACR classification
* Any extra-renal flare with an SLEDAI>6 and/or one BILAG A or 2 B
* Oral corticosteroids>10 mg/day and HCQ > 400 mg/day for at least 30 days prior to inclusion

Exclusion Criteria:

* Presence of active renal disease
* Previous intolerance or hypersensibility to any of the active components
* Active infection
* Unmeasurable levels of TMPT
* Pregnancy
* Presence of a severe flare that requires other immunosuppressive treatment for its control
* Any Psychiatric or social condition that did not ensure the patient´s follow-up and patient´s collaboration
* Previous treatment with EC-MPS or Azathioprine in the last 2 months
* Previous treatment with biological therapy in the last 3 months for anti-TNF therapy or in the last year for anti-CD20 therapy
* ALT or GPT >120 UI/mL non-lupus related in the last 30 days
* Leucopenia <1000x10E6 non-lupus related in the last 30 days
* Symptoms related to other medical conditions non-lupus related such as antiphospholipid syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Obtention of complete remission | 24 months
  Complete remission will be defined by a SLEDAI<4 and/or absence of any BILAG A or B after 12 weeks of treatment

SECONDARY OUTCOMES:
To evaluate the safety, improvement in biological parameters and reduction of number of extra-renal flares. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP ORDI-ROS, MD, Study Director — VALL D'HEBRON HOSPITAL; JOSEFINA CORTES HERNANDEZ, MD, Principal Investigator — VALL D'HEBRON HOSPITAL
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Ordi-Ros J, Saez-Comet L, Perez-Conesa M, Vidal X, Mitjavila F, Castro Salomo A, Cuquet Pedragosa J, Ortiz-Santamaria V, Mauri Plana M, Cortes-Hernandez J. Enteric-coated mycophenolate sodium versus azathioprine in patients with active systemic lupus erythematosus: a randomised clinical trial. Ann Rheum Dis. 2017 Sep;76(9):1575-1582. doi: 10.1136/annrheumdis-2016-210882. Epub 2017 Apr 27. PMID 28450313